CLINICAL TRIAL: NCT02767960
Title: Change of Serum Tenascin-C Concentration and the Relationship With Hs-CRP，cTnI and Prognosis in Patients With Acute Coronary Syndrome
Brief Title: Serum Tenascin-C Concentration in Patients With Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, Rchuang, Professor, The First Affiliated Hospital of Dalian Medical University
Other Study IDs: LCKY2016
Record Dates: First submitted 2016-05-03; First posted 2016-05-11 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Acute Coronary Syndrome
Keywords: Tenascin-C
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- STEMI group: The study population consists of 30 patients with ST-elevated acute myocardial infarction (STEMI,n = 30) who are admitted within 24 hours after chest pain attack. They will all undergo coronary angiography. The diagnosis is made according to American Heart Association (AHA, 2014 and 2015) guidelines. Patients who had autoimmune diseases, malignancies, chronic or acute infections, asthma, severe heart failure (NYHA class 3 and 4) and advanced liver or renal diseases are excluded.
- NSTEMI group: The study population consists of 30 patients with non-ST elevated acute myocardial infarction (NSTEMI,n=30) who are admitted within 24 hours after chest pain attack. They will all undergo coronary angiography. The diagnosis is made according to American Heart Association (AHA, 2014 and 2015) guidelines. Patients who had autoimmune diseases, malignancies, chronic or acute infections, asthma, severe heart failure (NYHA class 3 and 4) and advanced liver or renal diseases are excluded.
- UAP group: The study population consists of 30 patients with unstable angina pectoris (UAP, n = 30). They will all undergo coronary angiography for the diagnosis of acute coronary syndrome. The diagnosis is made according to the criteria of the American Heart Association (AHA, 2014 and 2015). Patients who had autoimmune diseases, malignancies, chronic or acute infections, asthma, severe heart failure (NYHA class 3 and 4) and advanced liver or renal diseases are excluded.
- control group: 15 age and body mass index matched healthy subjects with neither coronary artery disease nor any of the components of the metabolic syndrome are studied as Normal group.

SUMMARY:
This study valuates the serum Tenascin-C concentration in patients with acute coronary syndrome.

DETAILED DESCRIPTION:
It is found that Tenascin-C plays an important role in ventricular remodeling, heart failure, aortic dissection, rheumatic heart disease and other cardiovascular diseases, which may be a new marker for the diagnosis and prognosis prediction of these diseases. However, there is few relevant studies about the Tenascin-C concentration in patients with acute coronary syndrome.This study valuates the serum Tenascin-C concentration in patients with acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

.diagnosed as acute coronary syndrome,including STEMI,non-STEMI,and UAP.

* with left ventricular ejection fraction（LVEF）>=45%
* written informed consents are obtained
* admitted within 24 hours after chest pain attacked

Exclusion Criteria:

* complicated with rheumatic heart disease, coronary arteritis, hypertrophic cardiomyopathy or dilated cardiomyopathy
* complicated with malignant tumor,the immune system diseases, blood system diseases, recently (within 2 weeks) taking glucocorticoid drugs, the use of immunosuppressive agents and cerebral infarction
* with acute or chronic infection, surgery or trauma in the last month
* secondary hypertension, severe liver dysfunction,severe renal insufficiency
* with abnormal thyroid function or allergy to iodine agent
* refusal to sign the informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute coronary syndrome,including STEMI,non-STEMI,and UAP patients.
Sampling Method: Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Serum Tenascin-C concentration | 12 months
  Serum Tenascin-C concentration in ng/ml

SECONDARY OUTCOMES:
Relationship between Tenascin-C and high sensitive C reaction protein (hs-CRP) concentration | 12 months
  With or without association between them
Relationship between Tenascin-C and Troponin-I (Tn-I) concentration | 12 months
  With or without association between them
MACEs during 12-month follow-up | 12 months
  All major adverse cardiac events( MACEs) including death, myocardial infarction, angina, heart failure are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Rongchong Huang, doctor, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tamaoki M, Imanaka-Yoshida K, Yokoyama K, Nishioka T, Inada H, Hiroe M, Sakakura T, Yoshida T. Tenascin-C regulates recruitment of myofibroblasts during tissue repair after myocardial injury. Am J Pathol. 2005 Jul;167(1):71-80. doi: 10.1016/S0002-9440(10)62954-9. PMID 15972953
- [Background] Sato A, Aonuma K, Imanaka-Yoshida K, Yoshida T, Isobe M, Kawase D, Kinoshita N, Yazaki Y, Hiroe M. Serum tenascin-C might be a novel predictor of left ventricular remodeling and prognosis after acute myocardial infarction. J Am Coll Cardiol. 2006 Jun 6;47(11):2319-25. doi: 10.1016/j.jacc.2006.03.033. Epub 2006 May 4. PMID 16750702
- [Background] Fujimoto N, Onishi K, Sato A, Terasaki F, Tsukada B, Nozato T, Yamada T, Imanaka-Yoshida K, Yoshida T, Ito M, Hiroe M. Incremental prognostic values of serum tenascin-C levels with blood B-type natriuretic peptide testing at discharge in patients with dilated cardiomyopathy and decompensated heart failure. J Card Fail. 2009 Dec;15(10):898-905. doi: 10.1016/j.cardfail.2009.06.443. Epub 2009 Aug 26. PMID 19944367
- [Background] Nozato T, Sato A, Hikita H, Takahashi A, Imanaka-Yoshida K, Yoshida T, Aonuma K, Hiroe M. Impact of serum tenascin-C on the aortic healing process during the chronic stage of type B acute aortic dissection. Int J Cardiol. 2015 Jul 15;191:97-9. doi: 10.1016/j.ijcard.2015.05.009. Epub 2015 May 6. No abstract available. PMID 25965612